CLINICAL TRIAL: NCT05224154
Title: Re-Connect Usability, Feasibility, Acceptability, and Preliminary Efficacy Testing
Brief Title: Re-Connect Application for Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO-2020-123
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation; Acceptability of Health Care; Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Smoking Cessation; Patient Acceptance of Health Care; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Aim 1 will use small focus groups and feedback sessions (n = 4-6) to gain insight into the acceptability and usability of Re-Connect. Up to 3 single-case design studies (n = 4/round) will then be conducted to get more extended use of the app in a real world context to get additional information about usability and acceptability of the app. Aim 2 will involve a 2-group (AC vs SC), pilot randomized control trial to test the feasibility, acceptability, and preliminary efficacy of Re-Connect.
Who Masked: Participant
Masking Description: Participants will be told how they can earn back access to their applications but they will not be told whether this is considered the active or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abstinent Contingent (AC) Re-Connect (Experimental): Participants in this group will be able to unblock highly desired, but non-essential (e.g., social networking, shopping, games) applications contingent on meeting goals for smoking abstinence, as verified by meeting carbon monoxide goals (CO<=6ppm).
  Interventions: Behavioral: Abstinent Contingent (AC) Re-Connect
- Submission Contingent (SC) Re-Connect (Active Comparator): Participants in this group will also be able to unblock their applications, but contingent on submitting CO samples and independent of meeting CO goals for smoking abstinence.
  Interventions: Behavioral: Submission Contingent (SC) Re-Connect

INTERVENTIONS:
Behavioral: Abstinent Contingent (AC) Re-Connect — Participants in this group will be able to unblock highly desired, but non-essential (e.g., social networking, shopping, games) applications contingent on meeting goals for smoking abstinence, as verified by meeting carbon monoxide goals (CO<=6ppm).
  Arms: Abstinent Contingent (AC) Re-Connect
Behavioral: Submission Contingent (SC) Re-Connect — Participants in this group will also be able to unblock their applications, but contingent on submitting CO samples and independent of meeting CO goals for smoking abstinence.
  Arms: Submission Contingent (SC) Re-Connect

SUMMARY:
This series of studies will explore the acceptability, feasibility, and preliminary efficacy of making access to smartphone applications contingent on objective evidence of smoking abstinence.

DETAILED DESCRIPTION:
Aim 1 will use small focus groups and feedback sessions (n = 4-6) to gain insight into the acceptability and usability of Re-Connect. Up to 3 single-case design studies (n = 4/round) will then be conducted to get more extended use of the app in a real world context to get additional information about usability and acceptability of the app. Aim 2 will involve a 2-group (AC vs SC), pilot randomized control trial to test the feasibility, acceptability, and preliminary efficacy of Re-Connect.

ELIGIBILITY:
Inclusion Criteria:

* individuals who report smoking at least 10 cigarettes per day for at least 2 years, -18 years of age or older
* do not have any health complications that might interfere with the study or require more intensive treatment (e.g., emphysema, chronic obstructive pulmonary disorder, asthma, lactose intolerance)
* report a strong desire to quit smoking (8 or higher on a 10-point Likert scale)
* has prior experience using a smartphone, speak English, and are literate, will be eligible for the study.

Exclusion Criteria:

* Individuals with mental health complications that are either un-managed or that have been managed for less than 6-months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Survey | through study completion, up to 12-weeks
  A survey that participants in Aim 1 usability testing will complete after testing out the Re-Connect application. Focus and feedback group participants, as well as single-case design participants, will complete this survey and a score of 75 or higher will be required before moving to the RCT in Aim 2.
Reconnect use (RCT, Aim 2) | 6-months
  Over the 6-month observation period we will track the how much and to what extent participants use Re-Connect and continue to submit CO samples.
Duration of Re-Connect Use (RCT, Aim 2) | 6-months
  Over the 6-month study we will track how long participants are engaged with using Re-Connect.
Acceptability (RCT, Aim 2) | 6-months
  At three time points we will have the participants complete a Treatment Acceptability Questionnaire to provide quantitative and qualitative feedback on their experience with using Re-Connect.
Percent negative carbon monoxide samples | 6-months
  We will compare the percentage of CO samples that meet the abstinence goals during the 6-month study.
7-day point prevalence of self-reported, and CO verified, smoking | 6-months
  Participants will provide self-reports and a CO sample to confirm smoking status throughout the 6-month study.

SECONDARY OUTCOMES:
Initial Acceptability | 1 day
  Individuals who respond to our advertisement for a smoking cessation intervention will be given information about Re-Connect and then they will be given the option of continuing to participate or discontinuing. Participants who discontinue will be asked why they are not interested to inform future versions of the intervention to make it more widely acceptable and therefore more likely to be adopted by a broader population.

OTHER OUTCOMES:
Smartphone Use Moderators | 6-months
  Exploratory analyses will be conducted on potential moderator variables (e.g., baseline time spent on phone, number of apps downloaded/used, types of apps used).

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Raiff, PhD, Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be shared if there is an appropriate need expressed by the investigator.